CLINICAL TRIAL: NCT00270907
Title: A Phase I Study of CT-2103 in Combination With Gemcitabine in Metastatic Breast Cancer
Brief Title: CT-2103 in Combination With Gemcitabine in Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0133
Record Dates: First submitted 2005-12-28; First posted 2005-12-29 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Breast Cancer; Breast Cancer
Keywords: Metastatic Breast Cancer; Breast Cancer; CT-2103; Gemcitabine; Xyotax; Gemzar
MeSH Terms: conditions — Breast Neoplasms | interventions — paclitaxel poliglumex; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT-2103 + Gemcitabine (Experimental): CT-2103 135 mg/m^2 intravenous (IV) on Day 1. Gemcitabine 1000 mg/m^2 IV on Day 1 and 8.
  Interventions: Drug: CT-2103; Drug: Gemcitabine

INTERVENTIONS:
Drug: CT-2103 — 135 mg/m^2 IV on Day 1.
  Other Names: Xyotax
Drug: Gemcitabine — 1000 mg/m^2 IV on Day 1 and 8.
  Other Names: Gemzar

SUMMARY:
The goal of this phase I clinical study is to find the highest safe dose of gemcitabine and CT-2103 that can be given in combination for the treatment of metastatic breast cancer. The safety and effectiveness of this combination will also be studied. This clinical trial will be offered to patients who are being considered for treatment with gemcitabine. Research lab samples and research biopsies will not be requested as part of this study.

DETAILED DESCRIPTION:
CT-2103 is a chemotherapy drug designed to deliver an active chemotherapy medication (paclitaxel) inside of tumor cells. Gemcitabine is FDA approved for the treatment of breast cancer.

Before you can start receiving drug on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam. You will have a CT scan of the chest and abdomen, a bone scan, and a chest x-ray performed to document the size and location of the tumor(s). Blood (about 2 tablespoons) will be drawn for routine tests. Women who are able to have children must have a negative blood-pregnancy test.

If you are found to be eligible to take part in this study, you will be assigned to a dose of CT-2103. Participants in this study will be enrolled in groups of 3. The first group will receive the lowest dose of CT-2103. Each new group of patients will receive a higher dose until the highest safe dose is found. The dose that you receive will depend on how many patients have received CT-2103 before you. You will only be assigned to one dose level, and you will stay at this same dose level for the entire study unless you have a serious side effect that requires the dose to be decreased or stopped. All participants will receive the same dose of gemcitabine, though it too may be lowered if severe side effects occur.

Both CT-2103 and gemcitabine are given through a vein. On the first day of your therapy (called 'Day 1'), you will receive a routinely given medication, ondansetron (Zofran), that will help decrease the risk of nausea. About 30 minutes later, CT-2103 will be given over 10-20 minutes followed by gemcitabine over 30 minutes.

One week later ('Day 8'), you will receive gemcitabine through the vein over about 30 minutes. You will return to see your doctor 3 weeks after your first dose of chemotherapy ('Day 21'), and then this pattern or cycle of treatment will be given again.

You will continue on therapy as long as the cancer is being controlled and you are not having unexpected or intolerable side effects. All chemotherapy will be given at M. D. Anderson.

You will have blood (about 2 tablespoons) collected once a week while you are on study to monitor the effects of chemotherapy on your bone marrow and liver and kidney function. You will see your doctor every 3 weeks to monitor how you are tolerating the therapy. At these visits, your doctor will discuss any symptoms you are having, and you will have a physical exam. If you are taking warfarin (Coumadin) you will need to have blood (about 1 tablespoon) collected three times a week to monitor you warfarin levels.

After each 6 weeks of chemotherapy, you will have repeat scans to evaluate the effects of the study drugs upon your cancer.

Once you have stopped taking therapy with CT-2103 and gemcitabine, you will be asked to return to see your physician in about 6 weeks to evaluate how you are doing and to find out if there has been any additional change in the cancer. You will have a complete medical history and physical exam. You will have a CT scan of the chest and abdomen, a bone scan, and a chest x-ray performed to document the size and location of the tumor(s).

This is an investigational study. Gemcitabine is FDA approved for the treatment of breast cancer when given in combination with paclitaxel. Gemcitabine will not be provided free of charge. CT-2103 is not yet FDA approved and will be provided free of charge during the study. Any laboratory testing that is not standard of care will be paid for by the supporting company. About 18 women will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed breast cancer that is either metastatic or unresectable.
2. Patients must have received anthracyclines as treatment of either early stage or metastatic breast cancer.
3. Previous taxane therapy is allowed.
4. Age >/= 18 years. There is limited data regarding the use of CT-2103 in children under 18 and they will be excluded from this combination dose finding study.
5. Eastern Cooperative Oncology Group (ECOG) performance status </= 2 (Karnofsky >/= 60%).
6. Measurable disease is not required.
7. Previous endocrine therapies are allowed but should be discontinued prior to initiation of therapy.
8. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with institutional policy.
9. The effects of CT-2103 on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Females of childbearing potential are defined as females who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 months.
10. Patients must have normal organ and marrow function as defined below: leukocytes >/= 3,000/ul; absolute neutrophil count >/= 1,500/ul; platelets >/= 100,000/ul; total bilirubin within normal institutional limits; aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) </= 2.5 * institutional upper limit of normal; creatinine within normal institutional limits or creatinine clearance >/= 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal; coagulation prothrombin time (PT) and Partial thromboplastin time (PTT) within normal limits unless patients are already anti-coagulated for other reasons (i.e., atrial fibrillation, etc.).
11. Patients with Her-2/neu positive tumors should have received prior trastuzumab if clinically appropriate.

Exclusion Criteria:

1. Patients with preexisting neuropathy >/= grade 2.
2. Patients may not be receiving any other investigational agents.
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to CT-2103, gemcitabine or other agents used in study. History of typical paclitaxel- or docetaxel-induced Grade 1-2 hypersensitivity reactions is permitted.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study.
7. Previous history of stem cell transplantation.
8. History of central nervous system metastases.
9. While there is no strict exclusion based upon previous number of therapies, patients who experienced grade 3 or 4 hematologic toxicity requiring the use of white blood count (WBC) growth factor support during their most recent chemotherapy prior to enrollment are excluded. Exceptions to this would include patients who received growth factor support as mandated by a clinical study, and/or patients who have been off all chemotherapy for at least 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of CT-2103 | 21 days
  MTD defined as the level of CT-2103 at which 2 out of 6 patients had dose limiting toxicity (DLT) where the primary DLT events of CT-2103 are uncomplicated neutropenia, febrile neutropenia, and/or grade 3 neuropathy. Assessments during the first cycle of therapy, where cycle is 21 days.

SECONDARY OUTCOMES:
Number of Participants with Response | 6 weeks following chemotherapy
  Evaluation of response in participants with measurable disease after each 6 weeks of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Green, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas (UT) MD Anderson Cancer Center official website — http://www.mdanderson.org